CLINICAL TRIAL: NCT05792878
Title: The Observational Study of COVID-19 Infection and Its Clinical Prognosis in Chronic Hepatitis B Patients With Antiviral Therapy
Brief Title: Study of COVID-19 Infection and Its Clinical Prognosis in Chronic Hepatitis B Patients With Antiviral Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Director of Department of Hepatology Division 2, Beijing Ditan Hospital, Capital Medical University, Beijing Ditan Hospital
Other Study IDs: DTXY26
Record Dates: First submitted 2023-03-28; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Chronic Hepatitis B; COVID-19 Infection
Keywords: chronic hepatitis; COVID-19 infection; interferon
MeSH Terms: conditions — Hepatitis B, Chronic; COVID-19; Hepatitis, Chronic | interventions — Interferons; nas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interferon treatment group: Patients with chronic hepatitis B who received antiviral treatment with Interferon at the Second Department of Hepatology, Beijing Ditan Hospital Affiliated to Capital Medical University from February 2022 to December 2023 were enrolled.
  Interventions: Drug: Interferon
- nucleoside analogues treatment group: Patients with chronic hepatitis B who received antiviral treatment with nucleoside analogues at the Second Department of Hepatology, Beijing Ditan Hospital Affiliated to Capital Medical University from February 2022 to December 2023 were enrolled
  Interventions: Drug: nucleoside analogues

INTERVENTIONS:
Drug: Interferon — The naive treated patients with chronic hepatitis B were given antiviral treatment with interferon according to their condition.
  Other Names: peg-interferon alpha
  Groups: Interferon treatment group
Drug: nucleoside analogues — The naive treated patients with chronic hepatitis B were given antiviral treatment with nucleoside analogues according to their condition.
  Other Names: NAs
  Groups: nucleoside analogues treatment group

SUMMARY:
This is a two-way (retrospective and prospective) study of COVID-19 infection in an observational cohort of patients with chronic hepatitis B treated with antiviral therapy. Patients with chronic hepatitis B who received anti-HBV treatment in the Second Department of Hepatology, Beijing Ditan Hospital Affiliated to Capital Medical University from February 2022 to December 2023 were enrolled. After enrollment, demographic data of patients, information on antiviral treatment of chronic hepatitis B, COVID-19 vaccination, COVID-19 infection and COVID-19 incidence and treatment from January 2022 to pre enrollment, and data on HBV virus and serology, clinical biochemistry, liver and lung imaging, COVID-19 nucleic acid and COVID-19 antibody examination of patients were collected. After enrollment, prospective anti-HBV treatment, HBV virology, clinical biochemistry, liver imaging and COVID-19 infection and morbidity were observed. The patients with COVID-19 infection during the prospective observation period were observed for COVID-19 infection, onset and treatment, including body temperature, clinical symptoms, signs, cardiac examination, pulmonary imaging, COVID-19, clinical biochemistry, disease severity, time of virus negative conversion, hospital stay and outcome. The influence of COVID-19 infection on liver disease and the influence of interferon anti-HBV treatment on COVID-19 infection, its pathogenesis and prognosis were studied.

DETAILED DESCRIPTION:
This is a two-way (retrospective+prospective) study of COVID-19 infection in an observational cohort of patients with chronic hepatitis B treated with antiviral therapy. Patients with chronic hepatitis B who received anti-HBV treatment in the Department of Hepatology Division 2, Beijing Ditan Hospital, Capital Medical University from February 2022 to December 2023 were enrolled. After enrollment, demographic data of patients, information on antiviral treatment of chronic hepatitis B, COVID-19 vaccination, COVID-19 infection and COVID-19 incidence and treatment from January 2022 to pre enrollment, and data on hepatitis B virus and serology, clinical biochemistry, liver and lung imaging, COVID-19 nucleic acid and COVID-19 antibody examination of patients were collected. After enrollment, prospective anti hepatitis B virus treatment, HBV virology, clinical biochemistry, liver imaging and COVID-19 infection and morbidity were observed. The patients with COVID-19 infection during the prospective observation period were observed for COVID-19 infection, onset and treatment, including body temperature, clinical symptoms, signs, cardiac examination, pulmonary imaging, COVID-19, clinical biochemistry, disease severity, time of virus negative conversion, hospital stay and outcome. The influence of COVID-19 infection on liver disease and the influence of interferon anti hepatitis B virus treatment on COVID-19 infection, its pathogenesis and prognosis were explored.

ELIGIBILITY:
Inclusion Criteria:

* 1) HBsAg positive for 6 months.
* 2) Patients undergoing initial or ongoing antiviral treatment.
* 3) HBeAg status and HBV DNA level are not limited.

Exclusion Criteria:

* 1) Patients with decompensated liver cirrhosis or previous decompensated liver cirrhosis.
* 2) At the same time, it is associated with other viral infections, such as hepatitis A virus, hepatitis C virus, hepatitis D virus, hepatitis E virus, HIV, etc. - 3) Accompanied with other serious physical and mental diseases, including uncontrolled primary kidney, heart, lung, vascular, nervous, digestive, severe metabolic diseases (such as uncontrolled hyperthyroidism, diabetes, serious complications, adrenal diseases, etc.), immunodeficiency disease, and accompanied with serious infection; History of active or suspected malignant tumors or malignant tumors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During 48 weeks of the prospective observation period, the treated patients continuously use the original treatment. After the initial treatment patients are enrolled, they receive antiviral treatment with interferon or nucleoside analogues according to the needs of the disease. During the treatment period, the corresponding virology, serology, clinical biochemistry and liver imaging examinations of hepatitis B antiviral treatment were carried out every 3-6 months.
  During COVID-19 infection, the patient shall be checked for clinical symptoms, clinical biochemistry, blood routine, pulmonary imaging, COVID-19 and antibodies, as well as other organs and functional indicators required by clinical needs.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The rate of COVID-19 infection. | 48 weeks after therapy
  The rate of chronic hepatitis B patients infected with COVID-19 after initial antiviral treatment.

SECONDARY OUTCOMES:
The rate of severe disease after COVID-19 infection. | 48 weeks after therapy
  The rate of severe disease after COVID-19 infection for chronic hepatitis B patients after initial antiviral treatment.
The hospitalization rate and duration of COVID-19. | 48 weeks after therapy
  The hospitalization rate and duration of COVID-19 for chronic hepatitis B patients after initial antiviral treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, Doctor, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Department of Hepatology Division 2, Beijing Ditan Hospital, Beijing, Beijing Municipality, China